CLINICAL TRIAL: NCT05998356
Title: Long-term Assessment of Balloon Eustachian Tuboplasty for Obstructive Eustachian Tube Disease: A Multicenter Single-blinded Randomized Controlled Study
Brief Title: Long-term Assessment of Balloon Eustachian Tuboplasty for Obstructive Eustachian Tube Disease
Acronym: LASt-BET
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RECHMPL22_0551
Record Dates: First submitted 2023-06-07; First posted 2023-08-18 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Eustachian Tube Dysfunction
Keywords: Eustachian tube; Balloon Eustachian Tuboplasty; Eustachian Tubal Score
MeSH Terms: interventions — Catheterization

STUDY DESIGN:
Intervention Model Description: Subjects randomly assigned to the intervention (experimental) group will benefit from BET, and subjects in the control group will undergo a Eustachian tube catheter insertion for probing and flushing the Eustachian tube but without dilation.
Who Masked: Participant, Outcomes Assessor
Masking Description: The subjects will be blinded to the treatment arm, while surgeons cannot be blinded for obvious reasons. The data collection from post-operative visits will be performed by assessors blinded to the inclusion arm to minimize possible biases.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (BET procedure) (Experimental): Subjects randomly assigned to the intervention group will benefit from BET procedure
  Interventions: Device: Balloon Eustachian Tuboplasty (BET) under general anesthesia.
- Control group (Placebo Comparator): Subjects from control group will undergo insertion of catheter for probing and flushing the Eustachian tube, the catheter won't be dilated
  Interventions: Device: Insertion of catheter for probing and flushing the Eustachian tube under general anesthesia

INTERVENTIONS:
Device: Balloon Eustachian Tuboplasty (BET) under general anesthesia. — Subjects will undergo general anesthesia with intubation. After retraction of the inferior turbinate using Naphazoline, the balloon will be inserted under optical control through the pharyngeal ostium of the Eustachian tube and inflated two times at a pressure of 10 bars as instructed by the manufacturer.
  Arms: Intervention group (BET procedure)
Device: Insertion of catheter for probing and flushing the Eustachian tube under general anesthesia — Participants in the control group will benefit from the insertion of a dedicated catheter, TubaClean, into the Eustachian tube during 2 minutes with gentle washing with saline solution, and then the catheter will be removed. This type of device is used to wash the Eustachian tube lumina during ear surgery. Thus, the procedure in the control group will be very close to the BET, except that no dilation will be performed. No Eustachian tube dilation will occur in this control group since the diameter of the catheter itself is not large enough to cause dilation. Eustachian tube catheterization is not per se a treatment of ETD but just of mucosal plugs, and the investigators expect no effect of this catheter insertion on the outcomes of the study. At the end of the procedure, subjects will have nasal dressings similar to the BET procedure to ensure the blinding of the study.
  Arms: Control group

SUMMARY:
To date, more than 130 000 Balloon Eustachian Tuboplasty (BET) procedures have been performed worldwide. This procedure is proposed in case of Obstructive Eustachian Tube Dysfunction (OETD) with or without chronic otitis media. However, the effectiveness of this procedure is still discussed amongst otolaryngologist. Most of studies,were open label prospective studies comparing Eustachian tube function before and after surgical treatment. A recent meta-analysis suggests that BET procedure improves postoperative Eustachian tube function, but high-level evidence is still lacking. In this project, the investigators propose to perform the first blinded randomized controlled trial procedure to assess the changes of Eustachian tube function after BET in a population of subjects with chronic OETD with or without chronic otitis. Prognosis factors of efficacy will be also investigated during the study.

DETAILED DESCRIPTION:
Obstructive Eustachian Tube Dysfunction (OETD) is a common medical condition whose prevalence is estimated to be 4.6% in the general population. Subjects suffering from OETD display various symptoms such as ear fullness, hearing loss, muffled hearing, pain, especially during pressure changes (airplane, diving, mountain experience…), tinnitus, ticking or popping sounds, autophony, or balance disorders. Failure to treat OETD can lead to chronic otitis media with cholesteatoma which is a severe medical condition requiring multiple surgeries and frequently associated with a permanent hearing loss and several major complications including meningitis, facial palsy and labyrinthitis. OETD medical management (pressure equalization device, in addition to medical treatment of rhinosinusitis and GERD) can be used in adults. However, high level evidence of effectiveness of such a treatment is still lacking and the success rates are unknown.

Surgical treatment such as grommets (tympanostomy tube) is only a temporary solution that might work in children, but is less effective in adults, requiring multiple surgeries during the patients lifetime for their repeated. Grommets are treating only the consequences but not the cause of OETD.

In 2010, the team of Prof. Sudhoff in Bielefeld, Germany, proposed for the first time the Balloon Dilatation of the Eustachian tube as an alternative treatment of OETD. To date, more than 75 000 Balloon Eustachian Tuboplasty (BET) procedures have been performed worldwide. However, the effectiveness of this procedure is still discussed amongst ENT physicians. Indeed, no blinded controlled randomized clinical trial was performed to address the effects of BET on Eustachian tube function. Only one randomized clinical trial using objective measures as outcomes was published so far and compared the effect of BET in addition to medical management versus medical management alone in an open label study. Knowing that the success rates of medical management are not clearly established and probably depend on the medical treatment used, the effect of the surgical procedure remains uncertain with this design of study. Another randomized controlled study used a quality-of-life questionnaire as main outcome measure 6 weeks after surgery. No objective assessment was performed as major outcome and follow-up was not sufficient for the main outcome measure. Most of published studies so far were open label prospective studies comparing Eustachian tube function before and after surgical treatment.

In this project, the investigators propose to perform the first blinded randomized controlled trial versus control procedure to assess the changes of Eustachian tube function after BET in a population of subjects with chronic OETD with or without chronic otitis, and after medical treatment failure. Prognosis factors of efficacy will be also investigated during the study. The control procedure will consist in the insertion of an Eustachian tube catheter, causing no dilation of the Eustachian tube. This procedure will allow to evaluate the effect of the balloon inflation itself on tubal function, compared to the insertion of catheter tube for probing and flushing in the Eustachian tube only. The literature reports very low rates of complication of BET surgery making this control procedure acceptable in terms of risks. The use of this type of control procedure is justified by the fact that no other reference treatment can be proposed as a reference group, and blinding the patient to the investigational arm is needed to ensure the methodological validity of the study.

Simplified study calender:

Visit 0: Selection Visit During this visit, investigators will inform patients of the study.

Visit 1: Inclusion Visit (14 days - 3 months after V0):

The subject consent will be obtained. Medical and demographic data will be collected and study examinations will be performed. Patients will be also received for an anesthesiology consultation and after randomized the in the intervention or the control group arm.

Visit 2: 2 days-3 months after V1 Intervention under general anaesthesia: ETD or control procedure.

Visit 3: 2 months (±15 days) after V2 Medical data collection and study examinations as well as ETDQ-7 questionary (Eustachian Tube Dysfunction Questionary).

Visit 4: Final Visit - 6 months (±15 days) after V2 Medical data collection and study examinations as well as ETDQ-7 questionary. End of the study for the participant.

Unscheduled visits If subject gets in contact with the site between regular visits due to acute disorders, an unscheduled visit will promptly be performed at the site. During this additional visit a physical examination, a systematic interview for recording of Adverse Event should be performed.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 85 years
* Clinical symptoms of OETD with Eustachian tubal score less or equal to 7/14
* Failure of well conducted medical treatment (GERD, allergy, rhinosinusitis) including pressure equalization device used for 1 month or more
* ASA score 1 or 2 (ASA : American Society of Anesthesiologists)

Exclusion Criteria:

* Palatal cleft
* Anatomical anomaly of pharyngeal Eustachian tube ostium on the treated side
* Medical history of nasopharyngeal radiotherapy
* Medical history of middle ear surgery (except myringotomy and/or tympanostomy tube)
* Eardrum perforation in the treated side
* Contraindication of general anesthesia, or major risk of general anesthesia including ASA scores of 3 and 4
* Major nasal obstruction ipsilateral to the Eustachian tube to treat
* Medical history of previous Eustachian Tube Dilation
* Pregnant or nursing woman, or in childbearing age and not willing to use contraception
* Inclusion in another interventional clinical trial
* Protected and vulnerable adult
* Not covered by Health insurance
* Refusal to sign informed consent form
* Subjects unable to attend all scheduled visits or to comply with all trial procedures

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Eustachian Tubal Score (ETS) | ETS is calculated at the inclusion, between 2 and 5 months after the inclusion, and between 6 and 9 months after the inclusion
  The changes of Eustachian tube function will be addressed by the calculation of the difference between final (v4) and initial (v1) Eustachian Tubal Score (ETS). The ETS score is a composite score considering objective measures (tubomanometry, tympanic impedancemetry) and subjective measures (Valsalva maneuver efficacy, opening of the Eustachian tube).ETS score is highly correlated to tubal function.

SECONDARY OUTCOMES:
Tympanic impedancemetry | The measurement is performed at the inclusion, between 2 and 5 months after the inclusion, and between 6 and 9 months after the inclusion
  Tympanic impedancemetry will classify ear impedancetry as normal (A) or abnormal (B or C type curves)
Specific Eustachian tube dysfunction score | The ETDQ-7 questionnary is performed at the inclusion, between 2 and 5 months after the inclusion, and between 6 and 9 months after the inclusion
  Specific Eustachian tube dysfunction score will be assessed by the ETDQ-7 questionary that has been shown to be sensitive and specific for Eustachian tube diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Venail, MD, PhD, Principal Investigator — University hospital of Montpellier, FRANCE